CLINICAL TRIAL: NCT00719017
Title: Upper Vaginectomy Versus Brachytherapy in Patients With Early Stage Endometrial Cancer Treated With Laparoscopic Surgery: a Randomized Controlled Study.
Brief Title: Upper Vaginectomy Versus Brachytherapy in Patients With Early Stage Endometrial Cancer Treated With Laparoscopic Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Stefano Palomba, Associate Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03/2007
Record Dates: First submitted 2008-07-16; First posted 2008-07-21 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Early Stage Endometrial Cancer
Keywords: Brachytherapy; Early stage edometrial cancer; Quality of life; Recurrence; Treatment; Vaginectomy
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vaginectomy group (Experimental): Upper vaginectomy
  Interventions: Procedure: Upper vaginectomy
- Brachytherapy group (Experimental): Post-operative brachytherapy
  Interventions: Radiation: Post-operative brachytherapy
- Control group (Active Comparator): Standard treatment
  Interventions: Procedure: Standard procedures

INTERVENTIONS:
Procedure: Upper vaginectomy — Laparoscopic surgery with upper vaginectomy
  Arms: Vaginectomy group
Radiation: Post-operative brachytherapy — Laparoscopic surgery followed by brachytherapy
  Arms: Brachytherapy group
Procedure: Standard procedures — Laparoscopic surgery +/- brachytherapy +/- pelvic radiation
  Arms: Control group

SUMMARY:
Recent findings have suggested that laparoscopic surgery is safe and effective, as well as laparotomic one, for treating patients with early stage endometrial cancer (ESEC). Moreover, our long-term previous data have shown a trend in vaginal cuff recurrence in subjects who underwent laparoscopic approach to ESEC consisting of extrafascial hysterectomy, bilateral salpingo-oophorectomy, pelvic +/- para-aortic nodes dissections, regardless grading or lymphovascular space invasion.

Based on these considerations, the aim of the current protocol-study will be to compare two different strategies for vaginal cuff recurrences prevention in patients affected by ESEC treated with laparoscopic surgery. In particular, upper vaginectomy followed by observation will be compared to post-operative brachytherapy.

DETAILED DESCRIPTION:
Women with ESEC scheduled for laparoscopic surgery will be enrolled and randomized in three arms [vaginectomy group (VG), brachytherapy group (BG), and control group (CG)]. All laparoscopic procedures will consist of total hysterectomy, bilateral salpingo-oophorectomy, peritoneal washing, systematic inspection of peritoneal cavity and biopsy of each suspect lesion, and pelvic (and eventual para-aortic) lymphadenectomy. In VG an upper vaginecomy will be added to standard laparoscopic procedures followed by observation, whereas BG will receive post-operative brachytherapy. CG will be treated with standard protocol for management of ESEC according to National Comprehensive Cancer Network (www.nccn.org).

Safety and efficacy data will be recorded in each group for 24 months of follow-up.

Data will be analyzed using the intention-to-treat principle and a P value of 0.05 or less will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Early stage endometrial cancer

Exclusion Criteria:

* Other pre-malignancies and malignancies
* Major medical conditions
* Psychiatric disorders
* Current or past history of acute or chronic physical illness
* Premenstrual syndrome (PMS)
* Current or past (within 6 months from study enrolment) use of drugs influencing cognition, vigilance, and/or mood.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-09; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Vaginal cuff recurrences | 24 months

SECONDARY OUTCOMES:
Post-operative complications | six months
Adverse events | 24 months
Loco-regional recurrence rate | 24 months
Distant recurrence rate | 24 months
Quality of life | 24 months
Overall survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Department of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro; Fulvio Zullo, MD, Study Chair — Department of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro
Locations (1):
- "Pugliese" Hospital, Catanzaro, Italy

REFERENCES:
- [Background] Zullo F, Palomba S, Russo T, Falbo A, Costantino M, Tolino A, Zupi E, Tagliaferri P, Venuta S. A prospective randomized comparison between laparoscopic and laparotomic approaches in women with early stage endometrial cancer: a focus on the quality of life. Am J Obstet Gynecol. 2005 Oct;193(4):1344-52. doi: 10.1016/j.ajog.2005.02.131. PMID 16202724